CLINICAL TRIAL: NCT00844350
Title: The Effect of Oxytocin (OT) and Oxytocin Plus Human Chorionic Gonadotropin (hCG), in Cycles Induced by Letrozole or Clomiphene Citrate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tabriz University (Other)
Responsible Party: Manizhe sayyah melli, Tabriz university of medical scince
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8725
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2009-02-16 (Estimated); Status verified 2009-02

CONDITIONS: Ovarian Response
Keywords: Oxytocin; Letrozole; Induction of ovulation
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- letrozole+hCG (No Intervention)
  Interventions: Drug: letrozole , oxytocin,hCG,clomiphene citrate
- letrozole+oxytocin (No Intervention)
  Interventions: Drug: letrozole , oxytocin,hCG,clomiphene citrate
- letrozole+oxytocin+hCG (No Intervention)
  Interventions: Drug: letrozole , oxytocin,hCG,clomiphene citrate
- clomiphene citrate +oxytocin (No Intervention)
  Interventions: Drug: letrozole , oxytocin,hCG,clomiphene citrate
- clomiphene citrate +oxytocin+hCG (No Intervention)
  Interventions: Drug: letrozole , oxytocin,hCG,clomiphene citrate

INTERVENTIONS:
Drug: letrozole , oxytocin,hCG,clomiphene citrate

SUMMARY:
The specific aims of this study were to assess whether letrozole as an aromatase inhibitor plus hCG or OT alone, or in combination compared with CC, improves ovarian response.Ethical design of this study is based on the ethical guidelines of the Iranian Medical and Health Ministry which is accepted by Tabriz medical university ethical committee .

DETAILED DESCRIPTION:
In a randomized controlled prospective clinical study, a total of 177 infertile women with CC+hCG-resistant PCOS included. The candidates were selected for this study in the clinics of Tabriz University of Medical Sciences, East Azarbayejan Province, North West of Iran, from Oct. 2006 to Sep. 2007. Infertile women who had chronic anovulation and classical PCOS with CC+hCG failure were age <40 y , had patent tubes on hysterosalpingography, and no other pelvic pathology, participated in this study. The patients who had hypersensivity to any oxytocic medications, history of cardiovascular disease, and took anti-hypertensive medications were excluded. In addition, women with blood pressure less than 90/60 mmHg, abnormal spermogram, anxiety, excess prolactin levels, and other causes of infertility were excluded. All participants were given adequate information, and consent was obtained from each participant.

The candidates were randomly divided into five groups including; letrozole + hCG (36 patients) (group 1), letrozole + OT (35 patients) (group 2), letrozole +OT + hCG (35 patients) (group 3), CC + OT (35 patients) (group 4), and CC + OT + hCG (36 patients) (group 5). Participants received letrozole 2.5mg at first month and 5mg at the second and third month. Also, CC was used 50 mg at the first month, to 150 mg at the third month to stimulate follicular growth. Oxytocin (OXYTIP; manufactured by IPDIC, Rasht, Iran), 5 IU and hCG (Choriomon; manufactured by IBSA Institute Biochimique SA, CH-6903 Lugano), 5000 IU were also administrated to induce ovulation. All patients underwent transvaginal sonography on day 13 to document the numbers of follicles and endometrial thickness. Participants were evaluated for three courses of intervention. Oxytocin was injected intramuscularly after CC or letrozol stimulation had induced enlarged ovarian follicles ( >18 mm in diameter to 30 mm). Decision to give a 5 IU dose of OT was made according to the pilot study (30). The patients who had larger follicles (more than 30mm in diameter), were withdrawn. The patients, who achieved pregnancy at the first or second month, were also withdrawn. All participants were evaluated for the levels of plasma progesterone one week after the injection of OT, hCG, or combination of them. A follow-up visit was arranged for each group every month at the second day of menstruation until 3 months after recruitment or at any time during the trial if pregnancy was achieved.

ELIGIBILITY:
Inclusion Criteria:

* infertile women who had chronic anovulation
* classical PCOS with CC+hCG failure
* age <40 y
* had patent tubes on hysterosalpingography
* no other pelvic pathology
* participated in this study

Exclusion Criteria:

* hypersensitivity to any oxytocic medications
* history of cardiovascular disease
* took anti-hypertensive medications were excluded.
* women with blood pressure less than 90/60 mmHg
* abnormal spermogram
* anxiety
* excess prolactin levels
* other causes of infertility were excluded

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2006-10; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
number of follicles, endometrial thickness, and clinical pregnancy rate | first ,second and third month